CLINICAL TRIAL: NCT03338400
Title: Dexamethasone Administration To Improve Patient Recovery In Ambulatory Vaginal Reconstructive Surgery: Is There A Role?
Brief Title: Dexamethasone Administration To Improve Patient Recovery In Ambulatory Vaginal Prolapse Surgery: Is There A Role?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Eric Hurtado, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLA17028
Record Dates: First submitted 2017-10-20; First posted 2017-11-09 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Quality of Recovery; Same Day Surgery; Nausea and Vomiting, Postoperative; Vaginal Prolapse
Keywords: Quality of Recovery, Dexamethasone, Same day surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Uterine Prolapse | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Active Comparator): Patients in the Dexamethasone arm will be administered the drug at the time of induction.
  Interventions: Drug: Dexamethasone
- Normal Saline (Placebo Comparator): The placebo arm patients will receive normal saline at the time of induction.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — Patients will be randomized to Dexamethasone arm will receive 8mg (2ml) of Dexamethasone at the time of induction.
  Arms: Dexamethasone
Drug: Normal saline — Patients randomized to normal saline will receive 2ml of Normal saline at the time of induction.
  Arms: Normal Saline

SUMMARY:
To the investigators knowledge there are no studies in the literature evaluating the effect of Dexamethasone administration on patients undergoing outpatient vaginal prolapse surgeries.

DETAILED DESCRIPTION:
The lifetime risk of undergoing surgical intervention for pelvic organ prolapse (POP) is estimated to be 10% and it is projected that from 2010 to 2050, the number of surgeries for POP will rise by 47.2%, from 166,000 to 245,970. In 1980, accounting for the rising costs of health care, congress approved Medicare to reimburse procedures performed at outpatient and ambulatory surgery centers. This led to an increasing number of stress incontinence (SUI) procedures being performed in the ambulatory setting from 34,968 in 1996 to 105,656 in 2006. However, the number of ambulatory POP surgeries decreased in the same time period. This was possibly due to the increase in the mean age of women undergoing ambulatory procedures for POP and SUI during that time periods.

At the investigator's institution has performed outpatient surgeries for POP and SUI for the past 3 years. Patients have tolerated same day surgery with minimal complications. In the investigator's previous prospective study assessing satisfaction after outpatient surgeries for POP and SUI, patients had a decreased quality of recovery at 48 hours compared to baseline. The investigators also recognized that nausea and pain control could have been better addressed. Unpleasant postoperative nausea and vomiting, pain control, return to normal voiding and return of bowel function can influence the quality of recovery (QOR) from surgery.

Postoperative nausea and vomiting (PONV) and pain management are particularly troubling for the patients. This might also delay discharge and prolong convalescence from the surgery.

Several safe interventions have been assessed in the literature for alleviating PONV, pain and recovery from laparoscopic gynecologic surgery.

Dexamethasone is a potent corticosteroid that has been widely used for chemotherapy induced nausea and vomiting. The mechanism of action is not completely understood. It has been proposed that a single dose may hamper the production and release of anti-inflammatory mediators, thereby decreasing postoperative nausea, emesis, pain perception and Dexamethasone also has a central antiemetic effect by inhibition of prostaglandin and/or release of endogenous opioids. A recent metanalysis concluded that Dexamethasone administration at induction is safe.

Pauls et al in their recent study randomized patients undergoing vaginal prolapse surgery to receive Dexamethasone and noted a decrease in PONV and reduced requirement of a rescue antiemetic. Their model involved patients with overnight stay and the results may not be applicable to our population. They also noted that women who received Dexamethasone preoperatively were more likely to pass the voiding trial.

ELIGIBILITY:
Inclusion Criteria:

1. Women over the age of 18
2. Women scheduled for vaginal POP reconstructive surgery with or without concomitant anti-incontinence procedure and with or without hysterectomy
3. ASA class 1-2

Exclusion Criteria:

1. Daily use of steroids, antiemetics in the month prior to surgery
2. Chronic pain requiring daily opioid treatment
3. History of allergy/intolerance to Dexamethasone
4. ASA class 3
5. Numerical Pain score of more than 4 at baseline
6. Renal/Liver disease
7. Diabetes mellitus
8. Pregnancy
9. Inability to answer questionnaires
10. Any systemic infections
11. Immuno compromised status
12. Patients with planned overnight stay

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The surgeries that are performed are only vaginal prolapse surgeries in a female pelvic medicine and reconstructive surgery department.
Enrollment: 51 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Willy Davila, Principal Investigator — Department Head
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Normal Saline
Started | 25 | 26
Completed | 24 | 24
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Normal Saline | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 13 | 16 | 29
Age, Continuous [Mean (Full Range); unit: years] | 66 [40 to 83] | 65 [34 to 85] | 65 [34 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 20 | 22 | 42
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
Body Mass Index [Mean (Full Range); unit: kg/m2] | 26 [18 to 38] | 28 [21 to 39] | 27 [18 to 39]

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire: Quality of Recovery 40
Description: The primary aim is to evaluate whether standard administration of Dexamethasone at the time of anesthesia induction in patients undergoing vaginal reconstructive surgery would result in improved Quality of Recovery. The QoR-40 has 40 items that consider early postoperative health status of patients. These items cover five dimensions including emotional state (9 items), physical comfort (12 items), patient support (7 items), physical independence (5 items) and pain (7 items). All items are rated on a five-point Likert scale from one (worst) to five (best). All negative items were reversed to ease the interpretation. The total score (global score) was computed by summing all items. The minimum and maximum possible scores were 40 and 200, respectively.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone | Normal Saline
Number analyzed (Participants) | 24 | 24
score on a scale | 174 (14.49) | 167 (16.02)

2. Secondary Outcome: Nausea, Vomiting
Description: Clinically important nausea >50
Time Frame: 24 hrs
Population: patients with >50 on nausea scale
Measure: Number; unit: participants
Groups:
- Normal Saline; Dexamethasone: Postoperative nausea scale
Arm/Group | Normal Saline | Dexamethasone
Number analyzed (Participants) | 24 | 22
participants | 2 | 2

3. Secondary Outcome: Urinary Tract Infections
Description: Number of UTIs diagnosed in each group
Time Frame: until 6 weeks
Measure: Number; unit: participants
Groups:
- Normal Saline; Dexamethasone: Number of UTIs
Arm/Group | Normal Saline | Dexamethasone
Number analyzed (Participants) | 24 | 22
participants | 1 | 2

4. Secondary Outcome: Readmissions
Description: Any patient that is re-admitted to the hospital and the reason for re-admission will be collected.
Time Frame: 6 weeks
Population: Number or ER visits post-op
Measure: Number; unit: participants
Groups:
- Normal Saline; Dexamethasone: ER visits post-op
Arm/Group | Normal Saline | Dexamethasone
Number analyzed (Participants) | 24 | 22
participants | 4 | 1

5. Secondary Outcome: Pain Level
Description: numerical pain scale ranges from 0 to 10, where lower scores represent less pain.
Time Frame: 24 hours
Population: Pain score from 0-10
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Normal Saline; Dexamethasone: Postoperative pain scale
Arm/Group | Normal Saline | Dexamethasone
Number analyzed (Participants) | 24 | 22
score on a scale | 6.04 (2.8) | 4.77 (2.59)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 6 month period of time.
Arm/Group | Dexamethasone | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03338400/Prot_SAP_000.pdf